CLINICAL TRIAL: NCT02524717
Title: A Single-Dose, Open-Label Study to Evaluate the Pharmacokinetics of JNJ-56021927 in Subjects With Mild or Moderate Hepatic Impairment Compared With Subjects With Normal Hepatic Function
Brief Title: A Study to Evaluate the Pharmacokinetics of JNJ-56021927 in Participants With Mild or Moderate Hepatic Impairment Compared With Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107774; 56021927PCR1018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; JNJ-56021927

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- JNJ-56021927 (Experimental): Participants with mild and moderate hepatic impairment and with normal hepatic function will receive JNJ-56021927 240 milligram (mg) orally once on Day 1.
  Interventions: Drug: JNJ-56021927

INTERVENTIONS:
Drug: JNJ-56021927 — Participants will receive JNJ-56021927 240 milligram (mg) orally once on Day 1.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of JNJ-56021927 in participants with mild and moderate hepatic impairment.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-dose, single-center, non-randomized study of JNJ-56021927 in participants who either have hepatic impairment or qualify for the control group. The study consists of 3 Phases: Screening Phase (21 Days), open-label treatment Phase (8 Days) and follow up Phase (49 Days). The duration of participation in the study for each participant is approximately 78 Days. Primarily the pharmacokinetics of JNJ-56021927 will be measured. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinically stable hepatic function as confirmed by the serum bilirubin and transaminase levels measured during Screening and those measured within 24 hours prior to study drug administration
* Sign an informed consent document indicating that the participant understands the purpose of and procedures required for the study and are willing to participate in the study. Participants must not have hepatic encephalopathy greater than or equal to (>=) Grade 3 where the participant lacks the capacity to provide informed consent as judged by the investigator. Mild or moderate hepatic encephalopathy that would not impede informed consent in the investigator's judgment is permitted
* Willing and able to adhere to the prohibitions and restrictions as specified in the protocol
* If a man is sexually active with a woman of childbearing potential and has not had a vasectomy, he must agree to use an adequate contraception method as deemed appropriate by the Investigator, always use a condom during sexual intercourse, and agree to not donate sperm during the study and for 3 months after receiving the study drug
* Body mass index (BMI) between 18 and 35 kilogram (kg)/meter (m)^2 (inclusive), and body weight not less than 50 kg
* The participant must have a total Child-Pugh score of 5 to 6, inclusive (mild); or 7 to 9, inclusive (moderate); the investigator will determine hepatic impairment

Exclusion Criteria:

* Screening thyroid-stimulating hormone (TSH) level greater than (>) Upper Limit of Normal (ULN), or participants with known history of thyroid disorders
* Participant who is on thyroid replacement therapy
* History of drug abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 2 years before Screening or positive test result(s) for drugs of abuse (that is, opiates, barbiturates, benzodiazepines, cocaine, cannabinoids, and amphetamines) at Screening or Day -1. A positive test for participants with prescriptions for drugs that may interfere with the drug screen (that is, opiates and benzodiazepines) may be allowed
* Known allergy to the study drug or any of the excipients of the formulation
* Intention to donate blood or blood products during the study or for 3 months after the administration of the study drug
* A man who plans to father a child while enrolled in the study or for 3 months after receiving the study drug
* Known history of seizure or condition that may predispose to seizure or on medication that lowers seizure threshold
* History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs
* Gall bladder (example, cholecystitis and cholelithiasis) or biliary tract disease
* Clinically significant renal laboratory findings including serum creatinine level greater than (>) 1.5 times ULN
* Inability to fast for 12 hours
* History of or current clinically significant medical illness
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The Cmax is the maximum observed plasma concentration of JNJ-56021927.
Maximum Plasma Concentration Corrected for Unbound Fraction (Cmax_unb) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The Cmax_unb is the maximum observed plasma concentration corrected for unbound fraction of JNJ-56021927.
Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The Tmax is the time to reach the maximum observed plasma concentration of JNJ-56021927.
Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC[0-24]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC(0-24hrs) is the area under the plasma concentration-time curve from 0 to 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve From 0 to 168 Hours (AUC[0-168]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC(0-168hrs) is the area under the plasma concentration-time curve from 0 to 168 hours post dosing.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC[0-last]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration Corrected for Unbound Fraction (AUC[last_unb]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC(last_unb) corrected for unbound fraction is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC (0-infinity) is the area under the plasma JNJ-56021927 concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma JNJ-56021927 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time Corrected for Unbound Fraction (AUC[infinity_unb]) Post Dose of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The AUC(infinity_unb) is the area under the plasma JNJ-56021927 concentration-time curve from time 0 to infinite time corrected for unbound fraction, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma JNJ-56021927 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Percentage of Area Under the Plasma Concentration-Time Curve Obtained by Extrapolation (%AUC[infinity,ex]) | Pre-dose up to 1344 hours post-dose
  The %AUC[infinity,ex] is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100, (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Terminal Half-life (t[1/2]) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Elimination Rate Constant (Lambda [z]) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The Lambda (z) determined by first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time of Last Measurable Plasma Concentration (Tlast) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  Time to last measurable plasma concentration is evaluated.
Total Apparent Clearance (CL/F) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The CL/F is defined as Dose/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) of JNJ-56021927 | Pre-dose up to 1344 hours post-dose
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Metabolite to Parent Drug Ratio for Maximum Observed Plasma Concentration (MPR Cmax) | Pre-dose up to 1344 hours post-dose
  The (MPR Cmax) is metabolite to parent drug ratio for maximum observed plasma concentration.
Metabolite to Parent Drug Ratio for Area Under the Plasma Concentration-Time Curve From Time 0 to Last Observed Quantifiable Concentration (MPR AUC[0-last]) | Pre-dose up to 1344 hours post-dose
  The MPR AUClast is metabolite to parent drug ratio for area under the plasma concentration-time curve from time 0 to last quantifiable concentration (AUC [0-last]).
Metabolite to Parent Drug Ratio for Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (MPR AUC [0-infinity]) | Pre-dose up to 1344 hours post-dose
  The MPR AUC [0-infinity] is metabolite to parent drug ratio for area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUC [0-infinity]).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (56 days after dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Knoxville, Tennessee
  - San Antonio, Texas

REFERENCES:
- See also: A Single-Dose, Open-Label Study to Evaluate the Pharmacokinetics of JNJ-56021927 in Subjects With Mild or Moderate Hepatic Impairment Compared With Subjects With Normal Hepatic Function — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107774&attachmentIdentifier=abd44e16-069f-4d81-a8a3-0136dcf9b48a&fileName=CR107774_CSR.pdf&versionIdentifier=